CLINICAL TRIAL: NCT04338464
Title: The Roshni Project Phase 3: Developing a Culturally Driven Approach to Enhancing the Mental Well-being of Young South Asian Women
Brief Title: The Roshni Project - Developing a Psychosocial Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Gursharan Virdee, Research Analyst, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 022/2019
Record Dates: First submitted 2020-03-20; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Mood Disorders
Keywords: Cultural Relevance; Cultural Adaptation; South Asian; Gender
MeSH Terms: conditions — Mood Disorders; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Behavioral: Psychosocial therapy for South Asian women experiencing mood disorders

INTERVENTIONS:
Behavioral: Psychosocial therapy for South Asian women experiencing mood disorders — The 12 week intervention has four major components:
  * Relational theory (Belgrave, 2002) & South Asian identity development (Inman et al., 2001). These foundational components focus on strengthening cultural identity through the exploration of values, navigation and reconciliation of two cultures.
  * Transdiagnostic treatment of mood disorders (Ehrenreich-May et al., 2017). This component will focus on skill building in the areas of emotion awareness, resilience, adaptability, self-compassion and healthy coping strategies (Farchione et al., 2012; Bilek & Ehrenriech-May, 2012; Ritschel, Noriel & Lindsay, 2015).
  * Psychoeducation on mental health, sexual health, and substance use.
  * Peer support is a critical component of the intervention and will be provided by the peer researcher on the team. Participants will have access to optional individual peer support for 30 minutes to one hour per week for the duration of the intervention, this can be in person or telephone support.

SUMMARY:
The mental health sector is being called upon to develop and implement interventions for youth that attend to gender, age and cultural diversity (Mental Health Commission of Canada, 2016). The proposed project outlines the development and feasibility testing of a culturally driven transdiagnostic psychosocial intervention for South Asian women aged 16-24 years. We will recruit 30 participants to complete the 12 week psychosocial intervention. Pre, midpoint and post evaluations will be completed to asses change in mental health, self esteem and values, and also qualitative feedback on participant experiences of the intervention.

ELIGIBILITY:
Inclusion criteria:

* aged 16-24 years
* identify as a woman
* ancestry connected to India, Pakistan, Bangladesh and Sri Lanka
* formal diagnosis of mood or anxiety disorder
* completed high-school in Canada
* reside in the Greater Toronto Area
* speak conversational English

Exclusion criteria:

• individuals with developmental disabilities and serious mental illness e.g. schizophrenia spectrum, bipolar and personality disorders.

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Self define as female
Enrollment: 30 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Depression, Anxiety & Stress Scale (Lovibond & Lovibond, 1995) | Change from baseline depression, anxiety and stress at 12 weeks
  The Depression, Anxiety & Stress Scale (Lovibond & Lovibond, 1995) is a 42 item scale questionnaire with a 4 point likert scale from 0 to 4 measuring across three domains of depression, anxiety and stress. Total scores range from 0-168, with higher scores indicating greater symptom severity.

SECONDARY OUTCOMES:
Emotion Regulation Questionnaire (Gross & John, 2003) | Change from baseline emotion regulation at 12 weeks
  Emotion Regulation Questionnaire (Gross & John, 2003) is a 10 item survey assessing emotion regulatory processes including subscales for cognitive reappraisal and expressive suppression. The survey has a 7 point likert scale ranging from 0 (strongly disagree) to 7 (strongly agree), with total range from 0-70 with higher scores indicating better emotion regulation.

OTHER OUTCOMES:
Rosenberg Self Esteem Scale (Rosenberg, 1965) | Change from baseline self esteem at 12 weeks
  Rosenberg Self Esteem Scale (Rosenberg, 1965) is a 10 item self report measure used globally to assess self esteem amongst young adults. Scores on a 4 point likert scale with total scores ranging from 0-40, with higher scores indicating high self esteem.
Connor-Davidson Resilience Scale (Campbell Sills & Stein, 2007) | Change from baseline resilience at 12 weeks
  Connor-Davidson Resilience Scale (Campbell Sills & Stein, 2007) is a 25-item self report form including key features of resilience found across cultures including self-efficacy, action oriented approach, viewing change or stress as a challenge or opportunity, recognizing limits to control, faith and past successes. Scores range from 0-4, with full range from 0-100, and higher scores reflecting greater resilience.
Culture and Identity Schedule (Bhugra et al., 1999) | Change from baseline cultural identity at 12 weeks
  Culture and Identity Schedule (Bhugra et al., 1999) is a 106 item survey which explores adherence to traditional cultural values amongst immigrant South Asians in high income contexts. Items are scored 0 indicating more Eurocentric values and 1 indicating alliance with South Asian values. Higher total scores reflect greater overall affiliation with South Asian culture and identity.
Cultural Values Conflict Scale for South Asian women (Inman et al., 2001) | Change from baseline cultural values conflict at 12 weeks
  Cultural Values Conflict Scale for South Asian women (Inman et al., 2001) measures cultural adjustment among North American South Asian women specifically in the areas of family relations, sex role expectations, dating and premarital practices, and marriage. This 40 item scales scored on a 6 point likert scale, with total range from 0-240 and higher overall scores indicating greater conflict.
World Health Organization Quality of Life Scale (WHOQOL-BREF) (Skevington, Lofty, O'Connell, 2004) | Change from baseline quality of life at 12 weeks
  World Health Organization Quality of Life Scale (WHOQOL-BREF) (Skevington, Lofty, O'Connell, 2004) is a 26 item cross culturally valid measure of quality of life. Scores range from 0-100 with higher scores indicating better quality of life.
Working Alliance Inventory (Horvath & Greenberg, 1989) | 12 weeks
  Working Alliance Inventory (Horvath & Greenberg, 1989) is a 36 item questionnaire that assesses the relationship between client and clinician, measuring working, therapeutic and helping alliance. Items are scored on a 7 point likert scale, with three 12-item sub scales measuring task, bond and goal.
Demographics | Baseline
  A detailed demographic profile will be developed including age, gender, ethnicity, sexual orientation/identity, religion, family composition, immigration history, mental health history, school and employment history, characteristics of neighbourhoods.
Service Use & Access | Baseline
  We will record participants use of services related to their mental health.
Service Use & Access | 6 weeks
  We will record participants use of services related to their mental health.
Service Use & Access | 12 weeks
  We will record participants use of services related to their mental health.
Qualitative Interviews | 6 weeks
  Mid-point interview (week 6): Participants will be asked about their experiences of the intervention including access to the group, content, facilitation and out of session practice.
Qualitative Interviews | 12 weeks
  Post-treatment interview (week 12): In this interview participants will be asked about their total experience of the intervention including access to the group, content, facilitation and out of session practice, perceived impacts, probing what aspects of the intervention were helpful and those that weren't as helpful, and thoughts about how we can improve the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gursharan Virdee, Doctorate, Principal Investigator — Centre for Addiction and Mental Health

IPD SHARING:
Plan to Share IPD: No